CLINICAL TRIAL: NCT01048190
Title: The Phase I Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains
Brief Title: The Clinical Trial Protocol for the Inactivated Poliomyelitis Vaccine Made From Sabin Strains
Acronym: IPV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government); National Institute for the Control of Pharmaceutical and Biological Products, China (Other)
Responsible Party: Liao Guoyang, PhD, Institute of Medical Biology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: imbcams-01; SFDA2007L02021 (Other: China state food and drug adminstration)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-08

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliomyelitis Vaccine; Sabin Strains; poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Infants I-1 (Experimental): Biological: Inactivated Poliomyelitis Vaccine (Sabin strains). Group I-1: 15 infants received 3 doses of formulation C vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Infants I-2 (Experimental): 15 infants received 3 doses of formulation B vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart;
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)
- Infant I-3 (Experimental): 15 infants received 3 doses of formulation A vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart.
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strains)

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — 15 infants received 3 doses of formulation C vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart.
  Other Names: Sabin IPV,lot No.20080303
  Arms: Infants I-1
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — 15 infants received 3 doses of formulation B vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart;
  Other Names: Sabin IPV, lot No.20080302
  Arms: Infants I-2
Biological: Inactivated Poliomyelitis Vaccine (Sabin strains) — 15 infants received 3 doses of formulation A vaccine and 15infants received 3 doses of placebo 3x0.5ml intramuscular injections, one month apart.
  Other Names: Sabin IPV, lot No.20080301
  Arms: Infant I-3

SUMMARY:
The purpose of this study is to evaluate the safety and the immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains by different does.

DETAILED DESCRIPTION:
The Sabin IPV was manufactured with poliovirus type1, 2, 3 Sabin strains and Vero cells by micro-carrier culture in 550 liter bioreactors. The virus suspension was harvested ,ultra-concentrated, purified and inactivated with formalin. Three formulations A,B,C of Sabin IPV were used, the DAg contents for A were type1 45,type2 64,type3 67.5 DU /0.5ml/per dose; for B 30,32,45 DU/0.5ml/per dose; for C 15,16,22.5 DU/0.5ml/per dose.

This is a randomized, double-blind, placebo control phase 1 clinical trial. Total 130 individuals were selected ,including adults (n=20), children(n= 20) and infants(n= 90). Adults were randomized to two groups A1(n=10) and A2(n=10).Group A1 received one dose of B ,one month later group A2 received one dose of A for safety observation. Children were randomized to two groups C1(n=10) and C2(n=10) and followed the same vaccination and safety observation procedures as adults. Infants were randomly allocated to three groups I-1,I-2,I-3 for safety and immunogenicity study. Group I-1 were vaccinated with three doses of C(n=15) or placebo (n=15) on day 0,30,60,serum samples were collected before and 30 days after dose 3 for detecting neutralization antibody. The same procedures were followed by GroupI-2 for B and group I-3 for A as groupI-1 with 30 days intermission.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age from 60 days to 60 years old;
* Routine blood assaying (white blood cell, red blood cell, hemoglobin), liver (alanine transaminase)and kidney(blood urea nitrogen) functions are normal before vaccination;
* Adults, parent(s) or guardians are able to understand and sign informed consent for participation;
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions;
* Infants no vaccinated with poliovaccine or other preventive biologicals in recent 7 days;
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Have medical record of participants or their family on allergy, convulsion, falling sickness, encephalopathy and psychopathy;
* Abnormal results of routine blood assaying (white blood cell, red blood cell, hemoglobin), liver (alanine transaminase)and kidney(blood urea nitrogen) functions before vaccination;
* Low platelet or bleeding disorder do not allow vaccination into the muscle;
* Have damaged or lower immunological function;
* Received blood, plasma or immunoglobulin treatment since birth;
* Have inborn abnormality, develop obstacles or clinical diagnostic serious chronic ( Down Syndrome, diabetes, sickle cell anemia or neural Guillain-Barre Syndrome ).

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of Inactivated Poliomyelitis Vaccine made from Sabin Strains by different does. | one year

SECONDARY OUTCOMES:
To evaluate the immunogenicity of Inactivated Poliomyelitis Vaccine made from Sabin Strains by different does. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Liao Guoyang, PhD, Principal Investigator — Institute of Medical Biology, Chinese Academy of Medical Sciences; Li Rongcheng, MD, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control; Li Changgui, PhD, Principal Investigator — National Institute for the Control of Pharmaceutical and Biological Products, China
Locations (1):
- Hezhou Center for Disease Prevention and Control, Hezhou, Guangxi, China